CLINICAL TRIAL: NCT03625180
Title: An Observational, Prospective, Multicentre Study of Patients With Outerbridge Grade III / IV Chondral and/or Osteochondral Defects of the Knee Treated With Nanofractured Autologous Matrix-induced Chondrogenesis
Brief Title: An Observational, Prospective Study of Patients With Chondral and/or Osteochondral Defects of the Knee Treated With NAMIC
Acronym: KNAMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jordi Villalba Modol (Other)
Responsible Party: Sponsor-Investigator, Jordi Villalba Modol, Doctor, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Other Study IDs: 2017584
Record Dates: First submitted 2018-07-10; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Chondral Defect; Osteochondral Defect
Keywords: nanofractured autologous matrix-induced chondrogenesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: NAMIC technique
  Interventions: Biological: NAMIC: nanofractured autologous matrix-induced chondrogenesis

INTERVENTIONS:
Biological: NAMIC: nanofractured autologous matrix-induced chondrogenesis — the NAMIC technique consists in: debridement of damaged tissue, removal of calcified cartilage with retention of healthy surrounding vertical cartilage, minimally invasive subchondral bone marrow stimulation, nanofracture (Nano FX, Arthrosurface, USA), and a posteriori protect the lesion, stabilization of the clot, and facilitate stem cell adhesion and proliferation that migrate from the bone marrow with a type I/ III collagen and elastine membrane (Cartimaix, Matricel, Germany).

SUMMARY:
It is a prospective observational study of hospital cases. The objective is to determine the decrease of lesion size and the regeneration of chondral tissue in femoral condyle cartilage defect treated with NAMIC.

24 patients will be included

DETAILED DESCRIPTION:
Background: The treatment of chondral lesions remains a challenge for orthopaedic surgeons. They are most common in young active individuals and result in substantial impairment of quality of life. The conventional joint treatment methods available to date, such as Pridie-type perforations, microfractures using open or arthroscopic approaches and mosaicoplasty are far from satisfactory. Cell-based therapies have also been tested in more advanced research centres.

Nanofractured autologous matrix-induced chondrogenesis (NAMIC) is a simple, easily reproducible implantation technique that can be performed in most hospitals to improve clinical outcomes of patients with severe chondral lesions.

The present observational, multicentre study is based on the recently published NAMIC© technique (Behrens_Bentin_06_2015 The Knee) that reports significant improvements over previous techniques, especially regarding the reduction of rehabilitation period. Our main aim is to confirm these results in a larger sample.

NAMIC is a matrix-guided minimally invasive stimulation of the subchondral bone marrow.

The present study will collect data on the usual medical practice when the NAMIC technique is used to treat grade III or IV symptomatic focal cartilage lesions.

According to Chen 2011 JOR 2011, nanofracture achieves a uniform blood drainage and pluripotential cell recruitment of the bone marrow through the depth of the 9mm perforations. As observed by Eldracher AJS 2014, it also allows a faster recovery thanks to the minimal aggression on the subchondral bone as the diameter of the drill holes is 1 mm.

According to the study published by Benthien JP, in Knee Surg Sports Traumatol Arthrosc 2011 Aug:19(8):1316-9, AMIC induces satisfactory chondrogenesis.

To date, the combination of nanofracture plus Cartimaix membrane has not been used in patients in our environment.

Hypothesis: The NAMIC technique is useful for the treatment of chondral lesions of the knee.

Objectives:

Main: Determine the decrease of lesion size and the regeneration of chondral tissue in femoral condyle cartilage defect treated with NAMIC.

Secondary: Assess the clinical results regarding pain, articular rigidity and function before surgery and 12 months postoperatively.

Description of technique: After localization of the chondral lesion, the NAMIC technique consists in: debridement of damaged tissue, removal of calcified cartilage with retention of healthy surrounding vertical cartilage, minimally invasive subchondral bone marrow stimulation, nanofracture (Nano FX, Arthrosurface, USA), and a posteriori protect the lesion, stabilization of the clot, and facilitate stem cell adhesion and proliferation that migrate from the bone marrow with a type I/ III collagen and elastine membrane (Cartimaix, Matricel, Germany).

Nanofracture is a subchondral bone perforation procedure using a 1mm-thick needle, with a depth of 9mm, 2mm apart , in a systemic spiral fashion in the whole periphery of the lesion, using a specially-designed kit (Nano FX, Arthrosurface, USA). It allows a reproducible, effective and minimally invasive stimulation of the subchondral bone. Nanofracture achieves a uniform blood drainage and pluripotential cell recruitment of the bone marrow through the depth of the 9mm perforations.

Subsequently, the lesion is traced with a template included in the kit (Cartimaix, Matricel, Germany), and the membrane is cut to the adequate size, bearing in mind that it expands 10% with hydration. The two-layer membrane is then implanted on the lesion, and left to be hydrated by the blood from the stimulated area (Image 2). Cartimaix is a two-sided type I/ III collagen and elastine membrane that includes a smooth side (intraarticular) and a rough side facing the cartilage. Finally, fibrin sealing is achieved (Tissel, Baxter, USA). This technique can be combined with a graft in osteochondral injuries, but these are not contemplated in the present study.

Variables:

Main variable: Amount of tissue repaired, calculating the filling area of the lesion. Magnetic resonance will be used to determine the filling area at 12-month outpatient follow-up visit.

The following information will be collected: a) size and localisation of the lesion; b) alignment determined by telemetry; c) surgeries of cartilage or that may directly or indirectly affect cartilage such as meniscectomy, osteotomy, microfracture, mosaicoplasty or ligament repair.

A series of intraoperative pictures will be collected.

Secondary variables:

Pain: Visual analogue scale (VAS) Function and articular rigidity: KOOS scale, Tegner Activity Scale during routine outpatients visits, at preoperative visit and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Outerbridge grade III or IV cartilage lesions localized in the medial or lateral condyle of the knee (Chondral lesions were diagnosed by magnetic resonance T2 mapping and graded according to the Outerbridge classification.).
2. Size of lesion between 1.5 cm2 and 6 cm2 (specify size, alignment, and telemetry)
3. Body mass index ≤ 30 kg/m2.
4. Age 18 to 50.
5. Stable or stabilized knee, with normal axis (<+/-5º)
6. The patients included in the study will accept to follow the recommended physiotherapy programme, including exercises to be performed at home.

Exclusion Criteria:

1. Any disease that, in the opinion of the investigator, may prevent the patient from completing the study or interfere with the assessment of the efficacy or security of the treatment proposed.
2. Patients with any disorder of coagulation of the blood or receiving anticoagulant therapy.
3. Patients with rheumatoid arthritis, bi- or tri-compartmental arthritis such as chondrocalcinosis and gout.
4. Malalignment of affected leg with valgus or varus > 5º (and/or > vs. contralateral leg)
5. Chondral lesion of the tibial plateau (mirror lesions).
6. Known allergy to metal (nitinol or stainless steel) and/or pork products.
7. Any general pathology that may not allow long-term data collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Outerbridge grade III or IV cartilage lesions localized in the medial or lateral condyle of the knee.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Amount of tissue repaired | 12 months
  Amount of tissue repaired, calculating the filling area of the lesion. Magnetic resonance will be used to determine the filling area at 12-month outpatient follow-up visit.

SECONDARY OUTCOMES:
Localisation of the lesion | preoperative, and at 12 months
  THe localisation of the lesion will be described, using magnetic resonance.
Size of the lesion | preoperative, and at 12 months
  Magnetic resonance will be used to determine the size of the lesion, measured in mm.
Mechanical alignment | preoperative, and at 12 months
  Limb alignment (anatomic relation of bone axes) determined by telemetry. Measured in degrees.
Surgeries of cartilage or that may directly or indirectly affect cartilage | 12 months
  Surgeries of cartilage or that may directly or indirectly affect cartilage such as meniscectomy, osteotomy, microfracture, mosaicoplasty or ligament repair
Pain in the knee: Visual Analogue Scale | preoperative, and at 12 months
  Pain measured with a Visual Analogue Scale (VAS), which is a self-reported, single question, 11 point scale (from 0 no pain, to 10 unbearable pain).
KOOS score | preoperative, and at 12 months
  KOOS (Knee injury and Osteoarthritis Outcome Score) is a self-reported measure including 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. KOOS subscale scores will be aggregated and averaged as the primary outcome.
Activity level: Tegner Activity Scale | preoperative, and at 12 months
  Patient's activity level measured with the Tegner Activity Scale (TAS). It is a self-reported measure including 11 levels of activity (from 0 to 10) measuring work and sport activities graded numerically.

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided